CLINICAL TRIAL: NCT02798367
Title: National, Phase II/III, Multicenter, Randomized, Double-blind, Controlled, Parallel,Effect of Melatonin 3mg and 5mg Plus Cognitive Behavioral Therapy for Insomnia (CBT-I) Compared to the CBT-I Alone in the Treatment of Insomnia Disorder
Brief Title: Melatonin 3mg and 5mg Compared to Cognitive Behavioral Therapy for Insomnia (CBT-I) in the Treatment of Insomnia
Acronym: Morfeu
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-MSZ-02-03(05/16)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Insomnia Disorder
Keywords: insomnia; cognitive behavioral therapy for insomnia; melatonin
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I plus Melatonin 3 mg (Experimental): It's a tablet manufactured by Aché S.A., composed of melatonin 3mg. Melatonin 3mg tablet will be dispensed to 65 participants (first stage) of this group in a cartridge of 3 blisters with 10 tablets each, totalizing 30 tablets. If this arm is the best set for the second stage, more 56 participants will be randomly allocated in this group.The participant shall administer 01 tablet orally every 24 hours one hour before bedtime. The duration of treatment may be 21(±2) days.
  CBT-I is a non-pharmacological effective treatment for insomnia disorder. Behavioral techniques of Sleep Hygiene and Stimuli control are the most used. The CBT-I guidelines are standardized in protocol.
  Interventions: Behavioral: CBT-I plus placebo; Drug: CBT-I plus Melatonin 3 mg
- CBT-I plus Melatonin 5 mg (Experimental): It's a tablet manufactured by Aché S.A., composed of melatonin 5mg. Melatonin 5mg tablet will be dispensed to 65 participants (first stage) of this group in a cartridge of 3 blisters with 10 tablets each, totalizing 30 tablets. If this arm is the best set for the second stage, more 56 participants will be randomly allocated in this group.The participant shall administer 01 tablet orally every 24 hours one hour before bedtime. The duration of treatment may be 21(±2) days.
  CBT-I is a non-pharmacological effective treatment for insomnia disorder. Behavioral techniques of Sleep Hygiene and Stimuli control are the most used. The CBT-I guidelines are standardized in protocol.
  Interventions: Behavioral: CBT-I plus placebo; Drug: CBT-I plus Melatonin 5 mg
- CBT-I plus placebo (Other): It's a tablet manufactured by Aché S.A,. composed of placebo. The participants shall administer the placebo tablets to enable the double-blind study. Placebo will be dispensed to 65 (first stage) and 56 (second stage) participants of this group and shall administer 01 tablet orally every 24 hours one hour before bedtime for 21(±2) days.
  Sleep hygiene is a psychoeducational intervention that teaches patients to prevent external or environmental factors generate adverse effects and harmful to sleep. The stimulus control technique is based on five instructions that encourages the patient to establish a proper sleep-wake rhythm and strengthens the links between the way for a quick and well consolidated sleep. The CBT-I guidelines are standardized in clinical protocol.
  Interventions: Behavioral: CBT-I plus placebo

INTERVENTIONS:
Behavioral: CBT-I plus placebo — Behavioral techniques of Sleep Hygiene and Stimulus Control standardized in clinical protocol plus placebo (01 tablet, orally, always at night one hour before bedtime) for 21(±2) days)
Drug: CBT-I plus Melatonin 3 mg — Behavioral techniques of Sleep Hygiene and Stimulus Control standardized in clinical protocol plus Melatonin 3 mg (01 tablet, orally, always at night one hour before bedtime) for 21(±2) days.
  Other Names: Melatonin
  Arms: CBT-I plus Melatonin 3 mg
Drug: CBT-I plus Melatonin 5 mg — Behavioral techniques of Sleep Hygiene and Stimulus Control standardized in clinical protocol plus Melatonin 5 mg (01 tablet, orally, always at night one hour before bedtime) for 21(±2) days.
  Other Names: Melatonin
  Arms: CBT-I plus Melatonin 5 mg

SUMMARY:
National clinical trials, phase II/III, combined in two stages, randomized, double-blind, controlled, parallel, study of superiority, in which three hundred and seven (307) participants of both sexes, aged equal or more than 55 years will be randomly allocated to one of three treatment groups. In the first stage. The group 01 will use Melatonin 3mg plus CBT-I, the group 02 will use Melatonin 5mg plus CBT-I and the group 03 will use CBT-I plus placebo.

Based on the results of an interim analysis will be making a decision on whether to proceed with the study and, if so, on which the doses will be selected for the second stage of the study, to be better studied. The final analysis of the treatments, melatonin in the selected dose plus CBT-I versus CBT-I alone and placebo, will include participants from both stages.

DETAILED DESCRIPTION:
The treatment of insomnia disorder can be accomplished through pharmacological and nonpharmacological approaches. Behavioral techniques of Sleep Hygiene and Stimuli control are the most used. The Sleep hygiene is a psychoeducational intervention that teaches patients to prevent external or environmental factors generate adverse effects and harmful to sleep. The stimulus control technique is based on five instructions that encourages the patient to establish a proper sleep-wake rhythm and strengthens the links between the way for a quick sleep and well established. Melatonin is a hormone that participates in the regulation of the sleep-wake cycle, which is produced and secreted primarily by the pineal gland in the dark period and prepares the individual to sleep. Melatonin is involved in the induction of sleep and has proven therapeutic action in insomnia disorders, and may also play a role in the circadian timing system of mammals and serve as a marker for "biological clock".

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria for insomnia disorder, according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition);
* Complaint of difficulty falling asleep;
* Ability to understand and consent their participation in this clinical study, expressed by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* Any finding of clinical/physical observation or laboratory examination to be interpreted by the investigator as a risk to the inclusion of the participant in the clinical study;
* Known hypersensitivity to drug components used during the study;
* Participant have any family relationship to the second degree or bond with employees or employees of Sponsor and Sites;
* Participant has used beta-blockers (in the last 30 days prior to screening visit), psychoactive drugs or sedative effect, such as, but not limited to: sedatives (in the last 14 days prior to screening visit), hypnotics (in the last 07 days prior to screening visit), muscle relaxants (in the last 11 days prior to screening visit), antihistamines first generation (in the last 08 days prior to screening visit), and antidepressants, antiepileptics, antipsychotics, among others (in the last 30 days prior to screening visit);
* Participants diagnosed with clinical diseases that interfere with sleep, such as chronic pain, nocturia, hypothyroidism, hyperthyroidism, severe heart disease, serious neurological and psychiatric disorders according to the assessment of the investigator;
* Participants diabetics insulin dependent;
* Sleep apnea moderate to severe - AHI > 20 (Apnoea-Hypopnoea Index) assessed by polysomnography at the baseline;
* Participants who work at night;
* Participant who has BMI ≥ 30;
* Participant score above 50 in Anxiety Inventory to assess the degree of anxiety;
* Participant with cognitive impairment, based on the result obtained in the Mini-Mental State Examination. The cognitive impairment will be considered with score below 13 points for illiterates, below 18 for participants with one to eight incomplete years of schooling, below 26 for those with education of eight or more years;
* Participant score above 20 on the Beck Inventory to assess depression;
* Abuse of alcohol or illicit drugs, according to the assessment of the investigator;
* Male participants who do not agree to use acceptable methods of contraception; 1) male participants: barrier methods, except surgically sterile (vasectomy) or participants who declare to perform sexual practices on a not to reproductive way. 2) methods of contraception for the male participant's partner: oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, hormonal patch, tubal ligation and barrier methods; except surgically sterile (bilateral oophorectomy or hysterectomy) or the menopausal for at least one year;
* Female participants who are in the reproductive age and do not agree to use acceptable methods of contraception (oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation); except surgically sterile (bilateral oophorectomy or hysterectomy), the menopausal for at least one year and participants who declare to perform sexual practices on a not to reproductive way;
* Women in gestation period or who are breastfeeding;
* Participant who has participated in clinical trial protocols in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to the same.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of Sleep Latency after 21 (±2) days of the treatment. | 21 (±2) days
  Absolute change in sleep latency (in minutes) at the end of treatment compared to baseline. Sleep latency will be assessed by polysomnography.

SECONDARY OUTCOMES:
Quality of Sleep - Pittsburgh Sleep Quality Index | 21 (±2) days
  Absolute change the overall score PSQI-BR, at the end of treatment from baseline
Wellness Day - Well-Being Index-5 (WHO-5) | 21 (±2) days
  Absolute change the overall score of the WHO-5 level, in the range of 0 to 100 points, at the end of treatment from baseline.
Severity of Insomnia - Insomnia Severity Index | 21 (±2) days
  Absolute change the overall score of the Insomnia Severity Index at the end of treatment from baseline
Total Sleep Time - Polysomnography | 21 (±2) days
  Evaluate the total sleep time by polysomnography at the end of treatment from baseline
Sleep Architecture - the length and proportion of N1(non-rapid eyes movement) stages, N2, N3 and REM | 21 (±2) days
  Proportion of participants with sleep architecture classified as normal or abnormal, assessed by polysomnography at the end of treatment from baseline.
Sleep Efficiency - Polysomnography | 21 (±2) days
  Sleep efficiency variation assessed by polysomnography at the end of treatment from baseline
The Latency of Persistent Sleep - Polysomnography | 21 (±2) days
  Latency of persistent sleep variation assessed by polysomnography at the end of treatment from baseline
Latency of REM (rapid eyes movement) Sleep - Polysomnography | 21 (±2) days
  Latency of REM sleep variation assessed by polysomnography at the end of treatment from baseline
Satisfaction of the participants with the treatment. | 21 (±2) days
  Proportion of participants in each level of satisfaction category Likert 5 point (1. totally dissatisfied, 2. dissatisfied, 3. neither satisfied nor dissatisfied, 4. satisfied, 5. completely satisfied) evaluated comparing the groups at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Crippa Jr., Principal Investigator — Allergisa Search Dermato Cosmetic Ltda.
Locations (8):
- Brazil (8):
  - CEDOES - Centro de Diagnóstico e Pesquisa da Osteoporose do Espirito Santo., Vitória, Espírito Santo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Allergisa Pesquisa Dermato Cosmética Ltda., Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto USP, Ribeirão Preto, São Paulo
  - Centro de Estudos Multidisciplinar CEPES da Faculdade de Medicina do ABC, Santo André, São Paulo
  - Dr Consulta Clinica Medica Ltda, São Paulo
  - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda., São Paulo
  - Centro de Desenvolvimento em Estudo Clínicos Brasil - CDEC Brasil, São Paulo